CLINICAL TRIAL: NCT02717533
Title: Blood Volume Analysis and Renal Outcomes in Hemodialysis
Status: Completed | Type: Observational
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Principal Investigator, David S. Goldfarb, M.D., MD, VA New York Harbor Healthcare System
Other Study IDs: 01249-B
Record Dates: First submitted 2015-02-04; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: End Stage Renal Failure on Dialysis; Actual Impaired Fluid Volume; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- blood volume: dry weight adjusted according to ideal blood volume obtained from absolute blood volume measurement (Daxor)
  Interventions: Other: dry weight adjustment

INTERVENTIONS:
Other: dry weight adjustment — dry weight change to match ideal blood volume obtained by blood volume measurement.

SUMMARY:
The objective of the proposed study is to demonstrate that serial blood volume analysis (BVA) using RI-BVA (BVA-100, Daxor, NY) can be used to guide changes in prescription of dry weight for hemodialysis patients. The knowledge of a patient's ideal BV and degree of hypervolemia using these measurements can be used to change the prescription of DW in an objective way instead of the current standard of practice, which is based on subjective prescription of dry weight. A first study was conducted to determine the rate of plasma volume (PV) re-expansion for each patient as a guide to rate of fluid removal (results published, refer to citations). A second study was conducted in order to assess the value of a BVA measurement in guiding prescription of clinical DW. A follow up BVA would then be done in order to check if patients were closer to ideal BV than prior to changing dry weight.

DETAILED DESCRIPTION:
In the first study the investigators demonstrated that BV measurement using BVA-100 is useful to determine absolute BV as well as changes in BV and correlates reasonably well with CLM-III measurements. Individual refilling ability can be determined as well. This may prove useful in prescribing and monitoring ultrafiltration rates, establishment of optimal BV in HD patients and reducing morbidity and mortality associated with chronic HD.

In the current study the investigators hypothesize that BVA can be used in the longer term to evaluate the adequacy of the current clinically estimated dry weight in dialysis patients and can be used to titrate EDW in order to improve overall volume status and decrease the incidence of blood volume misinterpretation. The investigators enrolled 12 eligible patients. Participants underwent post-hemodialysis blood volume analysis (BVA) as a baseline measurement. Based on their Blood Volume (BV) status, their prescribed estimated dry weight (EDW) was adjusted. After 3 to 6 months, participants underwent a repeat BV measurement. The investigators compared the second value to the first in order to judge whether an improvement in BV status occurred if the dry weight prescription was changed, or to judge stability if it was not.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years
* Primary diagnosis of either chronic or acute kidney disease
* Currently receiving HD treatment
* Thrice-weekly or twice-weekly HD schedule
* Treated with standard bicarbonate HD for at least the preceding 6 months

Exclusion Criteria:

* Pregnant women or nursing mothers
* Known hypersensitivity to iodine, eggs, albumin or any other component of the Volumex injection kit
* Current enrollment in another investigational treatment protocol for dialysis
* Kidney transplantation
* Malignancy requiring chemotherapy
* Unmeasurable blood pressure with a sphygmomanometer
* Active hematological disease
* Active gastrointestinal bleeding
* Severe malnutrition (predialysis serum albumin <2.6 g/dL)
* Persistent condition of intradialytic blood pressure instability (hypotensive episodes in >80% of regular dialysis sessions) within the previous one month period

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Serial measurements of absolute blood volume before and after a hemodialysis treatment to achieve the target DW at which post-HD BV equals ideal BV | 6 months
  To demonstrate that serial BVA using the Blood Volume Analyzer (BVA-100) can be used to guide changes in prescription of DW for HD patients in an objective way instead of the current standard of practice, which is based on subjective prescription of dry weight. The results obtained from this first study have been published (see references) and show good correlation with CLM-III measurements and can estimate individual refilling ability
Serial measurements of absolute blood volume 3-6 months apart to achieve the target DW at which post-HD BV equals ideal BV | 6 months
  To demonstrate that serial BVA using the Blood Volume Analyzer (BVA-100) can be used to guide changes in prescription of DW for HD patients in an objective way so that post-dialysis weight reaches the patient's true dry weight. The other main objective is to study the correlation between change in post-dialysis weights and change in BV status as determined by BVA. This outcome will be looked at for all patients and also in the subgroups of patients who had their dry weight changed according to initial BVA measurement and in patients whose dry weight was kept the same after the initial measurement

SECONDARY OUTCOMES:
Incidence of dialysis complications and BV as determined by BVA | 6 months
  Dialysis complications that are under investigation include intradialytic hypotension and cramps. The investigators compare the incidence of dialysis complications for patients across subgroups of BV status as determined by BVA. We will also compare the incidence of dialysis complication at baseline and at the second measurement
Change in BV as determined by Crit-Line Monitor and reaching ideal BV by BVA | 6 months
  For every patient the investigators record the relative change in BV as determined by Crit-line monitoring. The investigators compare the relative BV change in patients who are euvolemic by BVA to those who are considered to be volume depleted and to the ones that are volume overloaded

CONTACTS AND LOCATIONS:
Locations (1):
- New York Harbor VA Healthcare System Hemodialysis Unit, New York, New York, United States

REFERENCES:
- [Result] Puri S, Park JK, Modersitzki F, Goldfarb DS. Radioisotope blood volume measurement in hemodialysis patients. Hemodial Int. 2014 Apr;18(2):406-14. doi: 10.1111/hdi.12105. Epub 2013 Nov 22. PMID 24262029
- [Derived] Malha L, Fattah H, Modersitzki F, Goldfarb DS. Blood volume analysis as a guide for dry weight determination in chronic hemodialysis patients: a crossover study. BMC Nephrol. 2019 Feb 11;20(1):47. doi: 10.1186/s12882-019-1211-7. PMID 30744587